CLINICAL TRIAL: NCT02015156
Title: Phase 1, Double-Blind, Randomized, Parallel-Group, Single-Dose, 2-Arm, Safety Study Of PF-05280014 And Trastuzumab Sourced From The US Administered To Healthy Male Volunteers
Brief Title: A Study Evaluating The Safety Of PF-05280014 And Trastuzumab In Healthy Male Volunteers (REFLECTIONS B327-06)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: B3271006; REFLECTIONS B327-06
Record Dates: First submitted 2013-12-06; First posted 2013-12-19 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Trastuzumab; Healthy Male Volunteers; Single-Dose; Phase 1; Biosimilarity
MeSH Terms: interventions — PF-05280014; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-05280014 (Experimental)
  Interventions: Biological: PF-05280014
- Trastuzumab-US (Active Comparator)
  Interventions: Biological: Herceptin®

INTERVENTIONS:
Biological: PF-05280014 — Concentrate for solution for infusion, sterile vial 150 mg, single-dose 6 mg/kg administered as 90-minute infusion on Day 1
  Other Names: Trastuzumab-Pfizer
  Arms: PF-05280014
Biological: Herceptin® — Concentrate for solution for infusion, sterile vial 440 mg, single-dose 6 mg/kg administered as 90-minute infusion on Day 1
  Other Names: Trastuzumab-US
  Arms: Trastuzumab-US

SUMMARY:
This study is to prove that there is no difference in the number of healthy male volunteers that will experience pyrexia (i.e. fever with body temperature of 38°C or higher) within a 24 hour period after administration of a single dose of 6mg/kg of PF-05280014 or trastuzumab sourced from the United States (trastuzumab-US). The study will also compare the safety of both drugs.

DETAILED DESCRIPTION:
Safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg^m2; and a total body weight >50 kg (110 lbs).
* Left ventricular ejection fraction (LVEF) within the normal range as measured by echocardiogram (ECHO) within 8 weeks prior to randomization.
* Subjects who have previously been exposed to a biologic agent (other than a HER2 inhibitor) may enroll provided that at least 3 months have passed since the last administration of that drug.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Previous exposure to an anti-HER2 antibody.
* History of serious allergic or anaphylactic reaction to a therapeutic drug or benzyl alcohol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of body temperature greater than or equal to 38.0 degrees Celsius | within 24 hours

SECONDARY OUTCOMES:
Incidence of pyrexia | within 24 hours
Severity of pyrexia | within 24 hours
Timing of pyrexia | within 24 hours
Seriousness of pyrexia | within 24 hours
Relationship of study therapy to pyrexia | within 24 hours
Incidence of body temperature greater than or equal to 38.0°C and/or use of concomitant treatment associated with fever suppression | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3271006&StudyName=A%20Study%20Evaluating%20The%20Safety%20Of%20PF-05280014%20And%20Trastuzumab%20In%20Healthy%20Male%20Volunteers%20%28REFLECTIONS%20B327-06%29